CLINICAL TRIAL: NCT00276874
Title: Preventing Cocaine Relapse: Developing Pharmacotherapies
Brief Title: Aripiprazole to Reduce Cocaine Relapse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig Rush (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Craig Rush, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DA020429; R01DA020429 (NIH); DPMC
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Addiction; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Experimental): Subjects receive oral aripiprazole.
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): Subjects receive oral placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole; 0-30 mg; oral; daily
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Placebos — Placebo; 0 mg; oral; daily
  Arms: Placebo

SUMMARY:
Despite the many behavioral and cognitive treatment therapies that exist for cocaine addiction, individuals who complete cocaine abuse treatment are still at high risk for relapsing. Aripiprazole, a medication that is currently used to treat schizophrenia, may be useful in preventing drug relapse in individuals addicted to cocaine. This three-part study will evaluate the interaction between aripiprazole and cocaine. It will also determine the safety and effectiveness of aripiprazole in preventing drug relapse among cocaine addicts.

DETAILED DESCRIPTION:
Cocaine addiction is a serious health problem with no available medical treatment for preventing relapse. Cocaine abusers often report that upon attempting to demonstrate control over the drug by only "sampling" it following a period of abstinence, they are more likely to relapse. These small "sampling" amounts of cocaine are thought to function as priming doses. Priming doses act as a stimulus in the brain to signal that there is more cocaine available, which in turn may lead to further cocaine use. Medications that reduce the stimulating effect of the cocaine priming dose may be useful in preventing cocaine relapse. Aripiprazole, a medication that is currently used to treat schizophrenia, may be effective at reducing relapse in individuals addicted to cocaine. By enhancing activity of the brain chemicals dopamine and serotonin, aripiprazole may counter the effects of cocaine and also reduce cocaine cravings.

This study will involve three sequential experiments. Experiment 1 will evaluate the physiological and behavioral effects of various combinations of cocaine and aripiprazole. Experiment 2 will evaluate the capability of aripiprazole at reducing the stimulating effects of cocaine. Lastly, Experiment 3 will evaluate the role of cocaine priming doses on subsequent cocaine use and how aripiprazole might alter the effect of the priming dose. In turn, these findings may lead to future clinical trials using aripiprazole to treat cocaine addiction and prevent relapse.

All three experiments will involve inpatient hospital stays. Participants will be required to refrain from using any non-study drugs, other than nicotine, and will undergo daily urine and breathalyzer tests. Questionnaires will be used to assess drug effects and cocaine cravings, and a computerized test will measure motor function and performance. Heart rate and blood pressure will be monitored periodically; an electrocardiogram (ECG) will record continuously to monitor heart electrical activity. Following the end of each experiment, all participants will be offered a referral to a drug abuse treatment program.

The first experiment will last 9 weeks and will enroll 8 individuals addicted to cocaine. Participants will take part in daily sessions in which they will receive varying doses of cocaine and aripiprazole, alone and in combination. This will provide important information regarding the safety and tolerability of cocaine-aripiprazole combinations.

The second experiment will last 10 weeks and will enroll 12 individuals addicted to cocaine. Participants will take part in various phases, which will each last several days. The phases will include a cocaine sampling phase; a cocaine acquisition phase in which participants will receive monetary rewards for distinguishing between cocaine and placebo; a placebo phase; an aripiprazole maintenance phase; a cocaine dose response phase in which the ability of aripiprazole to reduce cocaine's stimulating effects will be examined; and a washout phase in which no drugs will be given. Cocaine and aripiprazole doses will be determined by the results of the first experiment.

The third experiment will last 8 weeks and will enroll 12 individuals addicted to cocaine. A self-administration procedure designed to model relapse will be used to assess the effects of priming doses of cocaine on subsequent cocaine-taking behavior, alone and following aripiprazole treatment. Participants will be assigned to receive placebo for the first part of the study followed by aripiprazole for the remainder of the study or vice versa. During experimental sessions, participants will receive a specified amount of cocaine, which will act as the priming dose. Next, participants will choose between receiving either another similar dose of cocaine or money. This will be followed by a washout phase and then several more sampling-choice sessions with differing amounts of cocaine. Cocaine and aripiprazole doses will be determined by the results of the first experiment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for cocaine dependence
* Current cocaine use at study entry, as determined by a urine screen
* Body Mass Index of less than 30
* ECG results within normal limits
* If female, willing to use contraception throughout the study

Exclusion Criteria:

* Meets DSM-IV diagnostic criteria for dependence on any drugs other than cocaine or nicotine
* Currently seeking treatment for substance abuse
* Current or past serious illness, including impaired heart function, seizures, head trauma, or central nervous system tumors
* A family history of heart disease or seizures
* Current or past psychiatric disorder, other than substance abuse
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Behavioral effects of cocaine | Measured throughout the study

SECONDARY OUTCOMES:
Heart rate; blood pressure; ECG | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Craig R. Rush, PhD, Principal Investigator — University of Kentucky; Paul E Glaser, MD, PhD, Principal Investigator — University of Kentucky; Lon R. Hays, MD, Principal Investigator — University of Kentucky; Joshua A. Lile, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States